CLINICAL TRIAL: NCT00255437
Title: A Phase III Study of the Safety and Efficacy of Ferumoxytol (Compared With Oral Iron) as an Iron Replacement Therapy in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: Ferumoxytol Versus Oral Iron in the Treatment of Anemia in Non-Dialysis Dependent Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62745-7
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2007-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferrosoferric Oxide; Iron

INTERVENTIONS:
Drug: ferumoxytol or oral iron

SUMMARY:
The study will evaluate the safety and efficacy of a new intravenously administered iron drug to treat anemia in patients with chronic kidney disease who are not on dialysis.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of intravenous (IV) ferumoxytol as compared to oral iron in the treatment of anemia in non-dialysis dependent CKD patients. Patients are randomized to receive either two doses of 510 mg of ferumoxytol within one week or 200 mg oral elemental iron daily for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years.
* Have chronic kidney disease per K/DOQI guidelines.
* No change in EPO status during study.
* Baseline hemoglobin of ≤ 11.0 g/dl.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Received another investigational drug or device within 30 days.
* Recent parenteral or oral iron therapy.
* Patients with active GI bleeding or acute bleeding within 4 weeks.
* Patients that have other causes of anemia.
* Major surgery within 30 days or anticipated or planned major surgery during the study.
* Patients whose EPO status changes while on study.
* Patients with active infections.
* Recent blood transfusions.
* Patients with any known allergies to iron products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304
Dates: Start 2004-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The mean change in hemoglobin from baseline.

SECONDARY OUTCOMES:
Change in iron indices.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Phoenix, Arizona
  - Tempe, Arizona
  - New Haven, Connecticut
  - Augusta, Georgia
  - Peoria, Illinois
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Columbus, Mississippi
  - Broken Bow, Nebraska
  - Greenville, South Carolina
  - Charlottesville, Virginia
  - Norfolk, Virginia

REFERENCES:
- [Background] Landry R, Jacobs PM, Davis R, Shenouda M, Bolton WK. Pharmacokinetic study of ferumoxytol: a new iron replacement therapy in normal subjects and hemodialysis patients. Am J Nephrol. 2005 Jul-Aug;25(4):400-10. doi: 10.1159/000087212. Epub 2005 Jul 28. PMID 16088081
- [Result] Fishbane S, Bolton WK, Winkelmayer WC, Strauss W, Li Z, Pereira BJ. Factors affecting response and tolerability to ferumoxytol in nondialysis chronic kidney disease patients. Clin Nephrol. 2012 Sep;78(3):181-8. doi: 10.5414/cn107397. PMID 22874106
- See also: National Kidney Foundation — http://www.kidney.org/index.cfm